CLINICAL TRIAL: NCT01484171
Title: HLA-mismatched Microtransplantation for High Risk Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MST-AML-307PLAH-ASH
Record Dates: First submitted 2011-12-01; First posted 2011-12-02 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; idarubicin; Microtransplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- idarubicin (Active Comparator): The patients will receive induction chemotherapy containing standard dose of idarubicin in combination with cytarabine.
  Interventions: Drug: idarubicin
- microtransplantation (Experimental): The patients will receive induction chemotherapy containing high dose of idarubicin in combination with cytarabine and follow by infusioning granulocyte colony-stimulating factor-mobilized HLA-mismatched donor peripheral blood stem cells
  Interventions: Biological: microtransplantation

INTERVENTIONS:
Drug: idarubicin — idarubicin 10-12 mg/m2 for three days
  Arms: idarubicin
Biological: microtransplantation — idarubicin 10-12mg/m2 for four days. After chemotherapy infusion granulocyte colony-stimulating factor-mobilized HLA-mismatched donor peripheral blood stem cells following each of three cycles of high dose cytarabine chemotherapy
  Arms: microtransplantation

SUMMARY:
To compare the antitumor efficacy and toxicity of Idarubicin and cytarabine in combination with or not with infusions of granulocyte colony-stimulating factor-mobilized HLA-mismatched donor peripheral blood stem cells in patients with newly diagnosed high-risk acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

1. Having signed informed consent
2. Diagnosis was based on the French-American-British (FAB) and WHO criteria.
3. Age ≥ 7 years old
4. Age < 60 years old

Exclusion Criteria:

1.Patients with a blast crisis of chronic myeloid leukemia or acute promyelocytic leukemia

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
complete remission | one year

SECONDARY OUTCOMES:
disease-free survival | three years
overall survival | three years

CONTACTS AND LOCATIONS:
Overall Officials: huisheng ai, M.D., Principal Investigator — The Affiliated Hospital of the Chinese Academy of Military Medical Science
Locations (1):
- The Affiliated Hospital of the Chinese Academy of Military Medical Science, Beijing, Beijing Municipality, China